CLINICAL TRIAL: NCT03229499
Title: Pulmonary Hypertension and Anastrozole Trial (PHANTOM)
Brief Title: Pulmonary Hypertension and Anastrozole Trial
Acronym: PHANTOM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Johns Hopkins University (Other); University of Colorado, Denver (Other); Rhode Island Hospital (Other); Stanford University (Other); Vanderbilt University (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 827486; R01HL134905 (NIH)
Record Dates: First submitted 2017-07-18; First posted 2017-07-25 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Randomized Controlled Trial; clinical trial; anastrozole; pulmonary hypertension; pulmonary arterial hypertension; PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary | interventions — Anastrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Anastrozole (Experimental): 1mg (1 tablet)taken by mouth once a day for one year
  Interventions: Drug: Anastrozole
- Placebo (Placebo Comparator): 1 tablet taken by mouth once a day for one year
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Anastrozole — Anastrozole is an aromatase inhibitor indicated for:
  * adjuvant treatment of postmenopausal women with hormone receptor-positive breast cancer
  * first-line treatment of postmenopausal women with hormone receptor-positive or hormone receptor unknown locally advanced or metastatic breast cancer
  * treatment of advanced breast cancer in postmenopausal women with disease progression following tamoxifen therapy.
  Other Names: Arimidex
  Arms: Anastrozole
Drug: Placebo Oral Tablet — matching placebo tablet
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to determine whether the study drug, anastrozole may improve six minute walk distance at six months compared to placebo and to assess safety and side effects up to twelve months in pulmonary arterial hypertension (PAH).

ELIGIBILITY:
Inclusion Criteria:

* Previous documentation of mean pulmonary artery pressure > 25 mm Hg with a pulmonary capillary wedge pressure (or left ventricular end-diastolic pressure) < 16 mm Hg and PVR > 3 WU at any time before study entry.
* Diagnosis of PAH which is idiopathic, heritable, drug- or toxin-induced, or associated with connective tissue disease, congenital heart disease, portal hypertension, or HIV infection and receiving treatment for PAH.
* Most recent pulmonary function tests with FEV1/FVC >50% AND either a) total lung capacity > 70% predicted or b) total lung capacity between 60% and 70% predicted with no more than mild interstitial lung disease on computerized tomography scan of the chest.
* Ability to perform six minute walk testing without significant limitations in musculoskeletal function or coordination.
* If female, post-menopausal state, defined as:

  * > 50 years old and a) have not menstruated during the preceding 12 months or b) have follicle-stimulating hormone (FSH) levels (> 40 IU/L) or
  * < 50 years and FSH (> 40 IU/L) or
  * having had a bilateral oophorectomy.
* Informed consent.

Exclusion Criteria:

* Age < 18.
* Current treatment with estrogen, hormone therapy, or anti-hormone therapy (tamoxifen, fulvestrant, etc.)
* WHO Class IV functional status.
* History of invasive breast cancer.
* Clinically significant untreated sleep apnea.
* Left-sided valvular disease (more than moderate mitral valve stenosis or insufficiency or aortic stenosis or insufficiency), pulmonary artery or valve stenosis, or ejection fraction < 45% on most recent echocardiography (within 1 year).
* Initiation of PAH therapy (prostacyclin analogues, endothelin-1 receptor antagonists, phosphodiesterase-5 inhibitors, riociguat, selexipag) within three months of enrollment; the dose must be stable for at least three months prior to Baseline Visit. PAH therapy which is stopped and then restarted or has dose changes which are not related to initiation and uptitration will be allowed within 3 months prior to the Baseline Visit.
* Hospitalized or acutely ill.
* Renal failure (creatinine ≥ 2.0).
* Hypercalcemia.
* Severe osteoporosis: T score -2.5 to -3.4 without bone modifying treatment OR T score = - 3.5 or lower
* Child-Pugh Class C cirrhosis.
* Current or recent (< 3 months) chronic heavy alcohol consumption.
* Enrollment in a clinical trial or concurrent use of another investigational drug or device within 30 days of screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Kawut, MD, Principal Investigator — University of Pennsylvania
Locations (7):
- United States (7):
  - Stanford University, Stanford, California
  - University of Colorado - Denver, Aurora, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, East Providence, Rhode Island
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Derived] Kawut SM, Feng R, Ellenberg SS, Zamanian R, Bull T, Chakinala M, Mathai SC, Hemnes A, Lin G, Doyle M, Andrew R, MacLean M, Stasinopoulos I, Austin E, DeMichele A, Shou H, Minhas J, Song N, Moutchia J, Ventetuolo CE. Pulmonary Hypertension and Anastrozole (PHANTOM): A Randomized, Double-Blind, Placebo-Controlled Trial. Am J Respir Crit Care Med. 2024 Nov 1;210(9):1143-1151. doi: 10.1164/rccm.202402-0371OC. PMID 38747680

RESULTS

PARTICIPANT FLOW:
Groups:
- Anastrozole: 1mg (1 tablet)taken by mouth once a day for one year
  Anastrozole: Anastrozole is an aromatase inhibitor indicated for:
  * adjuvant treatment of postmenopausal women with hormone receptor-positive breast cancer
  * first-line treatment of postmenopausal women with hormone receptor-positive or hormone receptor unknown locally advanced or metastatic breast cancer
  * treatment of advanced breast cancer in postmenopausal women with disease progression following tamoxifen therapy.
Period: Overall Study
Arm/Group | Anastrozole | Placebo
Started | 43 | 41
Completed | 43 | 38
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anastrozole | Placebo | Total
Number analyzed (Participants) | 43 | 41 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (11.8) | 60.3 (10.2) | 59.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 17 | 16 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 41 | 36 | 77
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 31 | 33 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Six-minute walk distance [Mean (Standard Deviation); unit: meters] | 442.8 (119.5) | 416.3 (115.3) | 429.8 (117.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Six-minute Walk Distance
Description: Change in the distance walked in six minutes adjusted for baseline value and sex
Time Frame: 6 months
Population: Some participants are missing data at follow-up and the Analysis Population includes only participants with non-missing data. Includes non-missing six-minute walk distance at 6 months
Measure: Least Squares Mean (95% Confidence Interval); unit: meters
Arm/Group | Anastrozole | Placebo
Number analyzed (Participants) | 41 | 38
meters | 1.53 [-15.92 to 18.99] | 9.45 [-8.64 to 27.54]

2. Secondary Outcome: Change in Right Ventricular Function: Tricuspid Annular Systolic Plane Excursion (TAPSE)
Description: Change in tricuspid annular systolic plane excursion (TAPSE) adjusted for baseline value and sex. TAPSE is a measure of right ventricular function that is measured via cardiac echography
Time Frame: 6 months
Population: Some participants are missing data at follow-up and the Analysis Population includes only participants with non-missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Anastrozole | Placebo
Number analyzed (Participants) | 33 | 34
millimeters | -0.97 [-2.39 to 0.45] | -0.08 [-1.46 to 1.30]

3. Secondary Outcome: Change in Plasma NT-proBNP
Description: Change in log10 NT-proBNP adjusted for baseline value and sex
Time Frame: 6months
Population: Please note that some participants are missing data at follow-up and the Analysis Population includes only participants with non-missing data
Measure: Least Squares Mean (95% Confidence Interval); unit: log10(pg/ml)
Arm/Group | Anastrozole | Placebo
Number analyzed (Participants) | 40 | 39
log10(pg/ml) | 0.06 [-0.04 to 0.15] | 0.04 [-0.06 to 0.14]

4. Secondary Outcome: Change in the Medical Outcomes Study Questionnaire Short Form-36 (SF36) Physical Component Summary (PCS) Score Adjusted for Baseline Value and Sex.
Description: Change in the Medical Outcomes Study Questionnaire Short Form-36 (SF36) physical component summary (PCS) score adjusted for baseline value and sex. SF36 PCS score is a subjective measure of physical health status, with scores ranging from 0 to 100. Higher scores represent better health status.
Time Frame: 6months
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Anastrozole | Placebo
Number analyzed (Participants) | 42 | 40
units on a scale | 1.38 [-0.34 to 3.10] | 0.02 [-1.76 to 1.79]

5. Secondary Outcome: Change in the emPHasis-10 Score Adjusted for Baseline Value and Sex
Description: Change in the emPHasis-10 score adjusted for baseline value and sex. EmPHasis-10 is a pulmonary hypertension-specific measure of quality of life which is scored from 0-50, with higher scores indicating worse quality of life.
Time Frame: 6months
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Anastrozole | Placebo
Number analyzed (Participants) | 43 | 40
units on a scale | -0.27 [-2.34 to 1.81] | -0.51 [-2.68 to 1.66]

6. Secondary Outcome: Change in Actigraphy-measured Physical Activity: Change in 7-day Median Daily Vector Magnitude Count
Description: Actigraphy-measured vector magnitude count is an estimate of physical activity intensity. The total vector magnitude counts per day was measured over 7 days using an actigraphy device, and the median value over the 7 days was obtained. This outcome measure is the change in the 7-day median value from baseline to follow-up, adjusted for the baseline value, sex, and actigraphy device wear time.
Time Frame: 6months
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: counts per day(x10^5)
Arm/Group | Anastrozole | Placebo
Number analyzed (Participants) | 42 | 38
counts per day(x10^5) | -0.43 [-0.69 to -0.18] | -0.28 [-0.55 to 0]

7. Secondary Outcome: Number of Participants With a Clinical Worsening Event Between Anastrozole and Placebo Groups
Description: Number of participants with a clinical worsening event. Clinical worsening was defined as the addition of new PAH therapies or dose increases in previously stable PAH therapy for increased symptoms, hospitalization for PAH progression and/or right-sided heart failure, lung transplantation, atrial septostomy, or all-cause death.' Unit of Measure is retained as 'Participants.
Time Frame: 12 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Anastrozole | Placebo
Number analyzed (Participants) | 43 | 41
Participants | 7 | 8

8. Secondary Outcome: Change in Bone Mineral Density: Lumbar Spine Between Anastrozole and Placebo Groups
Description: Change in lumbar spine bone mineral density adjusted for baseline value and sex between anastrozole and placebo groups
Time Frame: 12 months
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: g/cm^2
Arm/Group | Anastrozole | Placebo
Number analyzed (Participants) | 43 | 34
g/cm^2 | 0 [-0.02 to 0.01] | 0 [-0.02 to 0.02]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Anastrozole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 3/41
Serious Adverse Events (participants affected / at risk) | 16/43 | 10/41
Other Adverse Events (participants affected / at risk) | 38/43 | 38/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anastrozole (N=43) | Placebo (N=41)
Catheter placement (Surgical and medical procedures) | 2 (2) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Heart Failure (Cardiac disorders) | 0 (0) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Carcinoma hepatocellular (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Chronic leg ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid retention in tissues (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Mallory Weiss tear (Gastrointestinal disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Pelvic mass (General disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subdural hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anastrozole (N=43) | Placebo (N=41)
Upper respiratory infection (Infections and infestations) | 9 (13) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (5)
Edema limbs (General disorders) | 5 (6) | 5 (5)
Hot flashes (Vascular disorders) | 6 (6) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (6)
Headache (Nervous system disorders) | 5 (8) | 4 (4)
Depression (Psychiatric disorders) | 3 (3) | 5 (5)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 2 (3)
Fatigue (General disorders) | 4 (6) | 3 (4)
Hypotension (Vascular disorders) | 2 (2) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Vaginal dryness (Reproductive system and breast disorders) | 2 (3) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 3 (3)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Palpitations (Cardiac disorders) | 0 (0) | 3 (3)
Presyncope (Nervous system disorders) | 0 (0) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT03229499/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT03229499/ICF_001.pdf